CLINICAL TRIAL: NCT03528915
Title: Conjunctivitis Incidence in the Newborn Within the First Week of Life: Impact of the Prophylactic Use of Rifamycine(CRY NOT).
Brief Title: Prevalence of Conjunctivitis and Indentification of Risk Factors With and Without Prophylactic Antibiotic Treatment in Neonates
Acronym: CRY-NOT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2014-34 Dr FONTAINE
Record Dates: First submitted 2018-04-19; First posted 2018-05-18 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Ophthalmia Neonatorum
Keywords: neonate, infant; eyewash; delivery room; prophylaxis; risk factor's
MeSH Terms: conditions — Ophthalmia Neonatorum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prophylaxis group: Newborns treated with rifamycin eye drops systemically two months before change of practices in delivery room.
  Interventions: Other: Rifamycine treatment
- no-antibiotic group: Newborns not treated with antibiotic prophylaxis in a systemic way, according to the new french guidelines of January 1st, 2015.
  Interventions: Other: whithout Rifamycine treatment

INTERVENTIONS:
Other: Rifamycine treatment — Phone prospecting: occurrence of conjunctivitis in newborns treated with rifamycine treatment in delivery room.
  Groups: Prophylaxis group
Other: whithout Rifamycine treatment — Phone prospecting: occurrence of conjunctivitis in newborns did not receive eye drop treatment in delivery room according to new guidelines.
  Groups: no-antibiotic group

SUMMARY:
The French guidelines for the use of Rifamycine eye drops in delivery room to prevent neonatal conjunctivitis have been actualized. Only newborns exposed to risk factors of conjunctivitis should be treated, compared to previous guidelines, treating all newborns. currently, there are no data describing risk factors for neonatal conjunctivitis. This study evaluated the incidence of conjunctivitis with or without Rifamycine eye drops treatment in the delivery room. Then risk factors for neonatal conjunctivitis where analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Newborns at the University Hospital of Amiens> 36SA,
* Admitted in maternity at the exit of nursery

Exclusion Criteria:

* Newborns at the Amiens University Hospital <36SA
* Eye drops for any medical reason within the first day of life.

Ages: 36 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns
Sampling Method: Non-Probability Sample
Enrollment: 881 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-07-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of conjunctivitis during the first 8 days of life in newborns | 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France